CLINICAL TRIAL: NCT02400632
Title: Assessment of the Novel MagicTouch Sirolimus Drug Coated Balloon Catheter for the Treatment of Coronary Lesions
Brief Title: MagicTouch Sirolimus Drug Coated Balloon Catheter for the Treatment of Coronary Lesions
Acronym: MAGIC-TOUCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAGIC TOUCH
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting balloon; in-stent restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MAGIC-TOUCH Drug-eluting balloon (Experimental): in-stent restenosis treated with drug-eluting balloon
  Interventions: Device: MAGIC-TOUCH Drug-eluting Balloon

INTERVENTIONS:
Device: MAGIC-TOUCH Drug-eluting Balloon — in-stent restenosis treated with drug eluting balloon

SUMMARY:
The purpose of this study is to demonstrate the efficacy of MagicTouch DCB in reducing late lumen loss / suppressing neointimal tissue formation as assessed by Quantitative Coronary Angiography / Intravascular Ultrasound examination for the treatment of coronary artery lesions ranging from 3.0 mm to 3.5 mm of diameter and lesion length ≤ 15 mm.

DETAILED DESCRIPTION:
Prospective, multicenter, randomized study designed to enroll 60 subjects with In-stent Restenosis, To demonstrate the efficacy of MagicTouch Drug-Coated Balloon in reducing late lumen loss / suppressing neointimal tissue formation as assessed by Quantitative Coronary Angiography / Intravascular Ultrasound examination for the treatment of coronary artery lesions ranging from 3.0 mm to 3.5 mm of diameter and lesion length ≤ 15 mm.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 and ≤ 80 years of age
2. Symptomatic ischemic heart disease;
3. Acceptable candidate for Coronary Artery Bypass Graft (CABG) or Angioplasty;
4. Target lesion located in a native coronary artery
5. Target lesion (maximum length is 15 mm by visual estimate) covered by a single balloon;
6. Reference vessel diameter must be ≥3.0 to ≤ 3.5 mm by visual estimate;
7. Target lesion ≥50% and <100% stenosed by visual estimate
8. Restenosis of initially stented main vessel.

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure;
2. Patient has had a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure;
3. Lesions in bypass grafts or bifurcations
4. Any non-target vessel or lesion intended to be treated during the index procedure, which is an unprotected left main, ostial lesion, chronic total occlusion (CTO), heavily calcified, bifurcation, vein grafts, have angiographic evidence of thrombus, be anything requiring atherectomy, thrombectomy, or pre-treatment with anything other than balloon angioplasty;
5. Patient presents with cardiogenic shock;
6. Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
7. Unprotected left main coronary artery disease with ≥50% stenosis;
8. Totally occluded target vessel (TIMI flow 0);
9. Calcified target lesion(s) which cannot be successfully pre-dilated;
10. A significant (>50%) stenosis proximal or distal to the target lesion that cannot be covered by same single balloon
11. Diffuse distal disease to target lesion with impaired runoff;
12. Left ventricular ejection fraction (LVEF) ≤30% (LVEF must be obtained within 1 months prior to the index procedure).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy assessed by the percentage (%) of in-stent neointimal tissue formation evaluated by Intravascular Ultrasound (IVUS) | 6-months after procedure

SECONDARY OUTCOMES:
Safety assessed by the composite rate for major adverse cardiac events at 12 months. (MACE: cardiac death, myocardial infarction (MI), target lesion revascularization (TLR) and Target vessel revascularization (TVR) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (3):
- Brazil (3):
  - Hospital Bandeirantes, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo